CLINICAL TRIAL: NCT03166345
Title: Use of Platelet Rich Plasma (PRP) for Improving Thin Endometrium For IVF Women
Brief Title: Use of Platelet Rich Plasma (PRP) for Improving Thin Endometrium
Acronym: PRPITM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Collaborators: Ganna Hospital (Other)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Lab Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Ibnsina-Ganna-PRP
Record Dates: First submitted 2017-05-18; First posted 2017-05-25 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Poor Endometrium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRP injection into Uterine Cavity (Experimental): PRP injection into Uterine Cavity For Treatment of Thin Endometrium
  Interventions: Other: Treatment of Thin Endometrium
- CSF (colony stimulating factor) (Experimental): CSF for Treatment of Thin Endometrium
  Interventions: Other: Treatment of Thin Endometrium
- No intervention (No Intervention): The control arm.

INTERVENTIONS:
Other: Treatment of Thin Endometrium — This is a trial to improve endometrial thickness by autologous injection of PRP into the Uterine Cavity compared with CSF or no treatment.
  Arms: CSF (colony stimulating factor); PRP injection into Uterine Cavity

SUMMARY:
Platelets rich plasma is simple source of growth factors and cytokines that can regulate endometrial growth for subgroup of thin endometrium women. It is an autologous source of this enhancing factors; therefore, there os no risk of using it within the same participant.

ELIGIBILITY:
Inclusion Criteria:

* women with thin endometrium

Exclusion Criteria:

* serum positive hepatitis B and C women

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Mean Diameter of endometrial thickness | 2 days
  How the endometrium would respond after 2 days of PRP

SECONDARY OUTCOMES:
Clinical pregnancy rate | 4 weeks or beyond after embryo Transfer
  Registered fetal heartbeat 4 weeks or beyond after embryo transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman S El-Gohary, MD, Principal Investigator — Ganna Hospital
Locations (2):
- Egypt (2):
  - Gannah IVF unit, Gannah Hospital, Giza
  - IbnSina IVF Center, IbnSina Hospital, Sohag

IPD SHARING:
Plan to Share IPD: No